CLINICAL TRIAL: NCT01060800
Title: The Genetics of Chiari Type I Malformation (CMI) With or Without Syringomyelia
Brief Title: The Genetics of Chiari Type I Malformation
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00011231
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2019-03

CONDITIONS: Chiari Type I Malformation
Keywords: Chiari; Chiari Type I; Chiari Type I Malformation; Familial Chiari
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duke University Medical Center is investigating the hereditary basis of Chiari type I malformations with or without syringomyelia (CM1/S). Our research is aimed at learning if CM1/S is indeed caused by factors inherited through the family and, if so, which genes are involved.

ELIGIBILITY:
The study is not currently enrolling new participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is not currently enrolling new participants.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-06; Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Genetic factors contributing to Chiari Type I malformation | end of study
  This study aims to identify genetic factors that contribute to or cause Chiari Type I malformation.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Ashley-Koch, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No